CLINICAL TRIAL: NCT01312350
Title: Concurrent Chemoradiation Versus Induction Docetaxel, Cisplatin and 5-fluorouracil (TPF) Followed by Concomitant Chemoradiotherapy in Locally Advanced Hypopharyngeal and Base of Tongue Cancer: A Randomized Phase II Study
Brief Title: Neoadjuvant Chemotherapy for Locally Advanced Squamous Cell Cancer of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-10-028
Record Dates: First submitted 2011-02-21; First posted 2011-03-10 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Hypopharyngeal Cancer
Keywords: neoadjuvant chemotherapy; definitive chemoradiation therapy; head and neck cancer; base of tongue; Locally advanced
MeSH Terms: conditions — Hypopharyngeal Neoplasms; Head and Neck Neoplasms | interventions — CF regimen; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCRT only arm (Active Comparator): no neoadjuvant chemotherapy before definitive CCRT
  Interventions: Drug: No treatment before definitive CCRT
- neoadjuvant chemotherapy arm (Experimental): 2 cycles of TPF chemotherapy before definitive CCRT
  Interventions: Drug: neoadjuvant docetaxel/cisplatin/fluorouracil

INTERVENTIONS:
Drug: neoadjuvant docetaxel/cisplatin/fluorouracil — 2 cycles of neoadjuvant Docetaxel/cisplatin/5-fluorouracil therapy followed by CCRT Neoadjuvant chemotherapy (docetaxel 75mg/m2 D1, cisplatin 75mg/m2 D1, 5-fluoruracil 759mg/m2/day, D1-4, every 3 weeks) CCRT protocol is same with that of control arm.
  Other Names: Docetaxel (taxotere)
  Arms: neoadjuvant chemotherapy arm
Drug: No treatment before definitive CCRT — concurrent chemoradiation therapy radiation: 70Gy/35fractions chemotherapy: cisplatin single 100mg/m2/day D1, D22, D43
  Arms: CCRT only arm

SUMMARY:
The investigators will examine whether 2-cycles of DFP chemotherapy before definitive concurrent chemoradiation therapy (CCRT) can improve progression-free survival in locally advanced (Stage III & IVM0) hypopharyngeal and base of tongue carcinoma compared to definitive CCRT alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven stage III/IVM0 hypopharyngeal or base of tongue cancer
* One or more evaluable or measurable lesion
* No prior chemotherapy, radiation, or surgery
* ECOG 0-2

Exclusion Criteria:

* Distant metastasis
* Other malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To determine whether addition of neoadjuvant chemotherapy before definite CCRT increase progression-free survival(PFS) compared with CCRT only | 18 months after the enrollment of the last patients

SECONDARY OUTCOMES:
To determine whether addtion of neoaduvant chemotherapy increase complete response rate compared with CCRT only | 18 months after enrollemnt of last patients
To determine whether addtion of neoaduvant chemotherapy increase organ preservation rate compared with CCRT only | 18 months after the enrollment of the last patient
To determine whether addition of neoadjuvant chemotherapy to CCRT increase the number of patients with adverse events compared with CCRT only | 18 months after the enrollment of the last patient

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea